CLINICAL TRIAL: NCT03292328
Title: Yoga for Chemotherapy-Induced Peripheral Neuropathy in Breast and GYN Cancer Survivors: A Pilot Study
Brief Title: Yoga for Symptoms of Nerve Damage Caused by Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-449
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Peripheral Neuropathy; Gynecologic Cancer
Keywords: breast cancer; neuropathy; peripheral neuropathy; yoga; 17-449
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Arm (Experimental): After randomization, participants in the Yoga group will meet twice weekly for 8 weeks of classes taught by MSK yoga instructors. Each class will last for sixty minutes. In addition to these group classes, participants will utilize a home-based program on the days group classes are not held. The daily home practice will continue for four weeks after the group classes are finished.
  Interventions: Other: Yoga
- Wait List Control Arm (WLC) (Active Comparator): Participants in the WLC group will continue usual care for twelve weeks before participating in Yoga classes for eight weeks. At the end of the twelve week follow-up, these participants will receive eight weeks of group Yoga classes and the home Yoga practice recording. At week 20, they will complete a final follow-up visit.
  Interventions: Other: Wait List Control

INTERVENTIONS:
Other: Yoga — Participants in the Yoga group will meet twice weekly for 8 weeks of classes taught by MSK yoga instructors. Each class will last for sixty minutes. In addition to these group classes, participants will utilize a home-based program on the days group classes are not held. The daily home practice will continue for four weeks after the group classes are finished.
  Arms: Yoga Arm
Other: Wait List Control — Participants in the WLC group will continue usual care for twelve weeks before participating in Yoga classes for eight weeks. At the end of the twelve week follow-up, these subjects will receive eight weeks of group Yoga classes and the home Yoga practice recording. At week 20, they will complete a final follow-up visit.
  Arms: Wait List Control Arm (WLC)

SUMMARY:
Some types of chemotherapy used to treat breast cancer can cause damage to nerves with symptoms like tingling, numbness, muscle weakness, and pain in the hands and feet that can last and can affect functioning. The purpose of this study is to find out the effects of yoga on reducing symptoms caused by such nerve damage.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age >/= 18 years old
* Survivors with a primary diagnosis of stage I-III breast, ovarian uterine, or endometrial cancer
* Moderate to severe chemotherapy induced peripheral neuropathy, defined by symptoms such as numbness, tingling, or pain ratings of 4 or greater on a 0-10 numeric rating scale
* Have completed neurotoxic chemotherapy, i.e. taxanes (paclitaxel, docetaxel) and platinum (carboplatin) at least 3 months prior to enrollment
* If taking anti-neuropathy medications, they are on a stable regiment (no change in 3 months)
* ECOG performance status 0-2

Exclusion Criteria:

* Participants with metastatic disease
* Participants who are currently receiving physical therapy or practicing yoga for any reason

Control Group - Inclusion/Exclusion Criteria

Inclusion Criteria:

* English speaking
* Age >/= 18 years old
* Survivors with a primary diagnosis of Stage I-III breast, ovarian, uterine, or endometrial cancer
* CIPN symptoms such as numbness, tingling, or pain ratings < 2 on a 0-10 NRS scale
* Have completed neurotoxic chemotherapy, i.e. taxanes (paclitaxel, docetaxel) and platinum (carboplatin) at least 3 months prior to enrollment
* ECOG performance status 0-2

Exclusion Criteria:

* Patients with metastatic disease
* Patients taking anti-neuropathy medication
* Patients who are currently receiving physical therapy or practicing yoga for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change in treatment related peripheral neuropathy symptoms | 8 weeks of the participants' most bothersome peripheral neuropathy symptom
  Treatment related symptoms will be evaluated by using NCI CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memoral Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhi WI, Baser RE, Zhi LM, Talukder D, Li QS, Paul T, Patterson C, Piulson L, Seluzicki C, Galantino ML, Bao T. Yoga for cancer survivors with chemotherapy-induced peripheral neuropathy: Health-related quality of life outcomes. Cancer Med. 2021 Aug;10(16):5456-5465. doi: 10.1002/cam4.4098. Epub 2021 Jul 2. PMID 34213086
- [Derived] Zhi WI, Chen P, Kwon A, Chen C, Harte SE, Piulson L, Li S, Patil S, Mao JJ, Bao T. Chemotherapy-induced peripheral neuropathy (CIPN) in breast cancer survivors: a comparison of patient-reported outcomes and quantitative sensory testing. Breast Cancer Res Treat. 2019 Dec;178(3):587-595. doi: 10.1007/s10549-019-05416-4. Epub 2019 Aug 27. PMID 31456070
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org